CLINICAL TRIAL: NCT00034632
Title: Open Label, Treatment Protocol for the Safety and Efficacy of Posaconazole (SCH 56592) in the Treatment of Invasive Fungal Infections
Brief Title: Study of Posaconazole in the Treatment of Invasive Fungal Infections (Study P02095)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P02095
Record Dates: First submitted 2002-05-01; First posted 2002-05-02 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Mycoses
Keywords: Aspergillosis, Candidiasis, Cryptococcosis, Phaeohyphomycosis; Invasive Fungal Infections
MeSH Terms: conditions — Mycoses; Aspergillosis; Candidiasis; Cryptococcosis; Phaeohyphomycosis; Invasive Fungal Infections

INTERVENTIONS:
Drug: Posaconazole oral suspension

SUMMARY:
This study is designed to evaluate the safety, tolerance and efficacy of Posaconazole (SCH 56592) under an open label, treatment protocol for subjects with invasive fungal infections:

A. which are refractory or resistant to standard antifungal therapies; B. for which there are currently no effective therapies; C. with a prior history of serious, severe or life-threatening toxicities while receiving antifungal therapy; D. with pre-existing organ dysfunction which precludes the administration of standard antifungal therapies.

DETAILED DESCRIPTION:
The current clinical trial is designed to provide posaconazole (SCH 56592 to subjects with invasive fungal infections a) which are refractory or resistant to standard antifungal therapies or b) for which there are currently no effective therapies. Subjects with such invasive fungal infections cannot be enrolled in controlled, randomized clinical trials. Secondly, this clinical trial is also designed to provide posaconazole (SCH 56592) to subjects with invasive fungal infections who c) have experienced serious or severe toxicities while receiving standard antifungal therapies or d) have pre-existing organ dysfunction such as renal dysfunction who require standard antifungal therapy which is precluded because of the toxicities associated with such therapy. This clinical trial also serves to allow collection of preliminary data regarding the safety and efficacy of posaconazole (SCH 56592) against a variety of invasive fungal infections which although serious and life-threatening are sufficiently rare so that they cannot be studied in a controlled, randomized clinical trial.

This is an open-label, treatment protocol for a multi-center study of posaconazole (SCH 56592) 200mg orally four times daily (QID) while hospitalized followed by posaconazole (SCH 56592) 400mg orally twice daily (BID) on discharge from hospital, in the treatment of invasive fungal infections. Approximately 320 subjects have been enrolled at 160 clinical study centers in the US and worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Proven or probable invasive fungal infections according to EORTC/MSG criteria.
* IFI are documented to be refractory to standard antifungal therapy OR intolerant to standard therapy.
* Able to take oral medication or take medication via enteral feeding tube.

Exclusion Criteria:

* History of serious or severe hypersensitivity or idiosyncratic reactions to azole antifungals.
* Concurrent progressive neurological disease (except if due to invasive fungal infection)
* Use of medications that are known to interact with azoles and that may lead to life-threatening side effects: terfenadine, cisapride, ebastine at entry or within 24 hours prior to therapy, or astemizole at entry or within 10 days prior to entry.concentration/efficacy of azole antifungals: rifampin, carbamazepine.
* Females pregnant or nursing.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-04; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

REFERENCES:
- [Result] Mezhir JJ, Mullane KM, Zarling J, Satoskar R, Pai RK, Roggin KK. Successful nonoperative management of gastrointestinal mucormycosis: novel therapy for invasive disease. Surg Infect (Larchmt). 2009 Oct;10(5):447-51. doi: 10.1089/sur.2008.049. PMID 19485785
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html